CLINICAL TRIAL: NCT01788514
Title: Combining Entertainment & Education Into an Age Appropriate Intervention Geared Toward Increasing Influenza Vaccination of Pediatric Patients in Underserved Communities
Brief Title: Combining Entertainment & Influenza Education for Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 11028
Record Dates: First submitted 2013-01-22; First posted 2013-02-11 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Videogame (Other): Subject will play educational videogame
  Interventions: Other: Videogame

INTERVENTIONS:
Other: Videogame — Subject will play an interactive educational videogame that is designed to increase their knowledge on influenza and the influenza vaccination.

SUMMARY:
The investigators have developed an influenza-vaccination-education-study-program that will involve the use of an animated influenza vaccine-based computer program (videogame) that is designed from the investigator's own initiative. The investigators propose implementing an influenza vaccination educational program in the pediatric satellite office that serves a population that has historical low rates of influenza vaccination.

DETAILED DESCRIPTION:
Each year, during the fall and winter, coinciding with the influenza season, the number of health care visits and the number of days missed from school increases due to febrile respiratory illnesses. The highest rates of influenza infections are present amongst school-age children. The vaccination against seasonal influenza remains the most important measure to prevent infection and to combat the overall spread of the virus. School-age children, in particular, adolescents, may not be aware of the need for influenza vaccination.

Interactive computerized educational programs have been developed and used in different pediatric settings in an attempt to increase children's understanding of their medical condition, and improve adherence to the treatment.

The investigators identified one of our satellite pediatric clinics, as being the perfect venue for an intervention that will attempt to increase influenza vaccination. The clinic is located in an underserved area. More than 9,000 children are seen annually in this clinic with about 20% of the patients age 8 and above. A pediatric pulmonary office, part of the pediatric clinic, serves a high number of patients, most of whom have poorly controlled asthma.

Currently, no focused, developmentally appropriate education programs regarding vaccination are used in our outpatient clinics.

The investigators propose implementing an influenza vaccination educational program in this pediatric satellite office that serves a population that has historical low rates of influenza vaccination.

The investigators have developed an influenza-vaccination-education-study-program that will involve the use of an animated influenza vaccine-based computer program (videogame) that is designed from the investigator's own initiative. This videogame should provide a basis or foundation to discuss the need for influenza vaccination and the adverse effects of influenza disease. It will be designed to intrigue the child by providing animated tours and creative experiences that are designed to encourage behavioral changes towards the need for vaccination.

The investigators hypothesis that by using this hybrid entertainment-educational tool, we will increase children's knowledge about influenza disease and the need for influenza vaccination. By using this age appropriate intervention, we aim to decrease children and adolescent's anxiety related to the vaccination and to increase vaccination rates. The investigators hypothesis that our intervention will have a high impact since it is geared to an ethnic community with historically low rates of influenza vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Children 8 years of age and older

Exclusion Criteria:

* Anyone who does not voluntarily give consent or assent to this study.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Increase the knowledge regarding influenza infection and influenza vaccination in school-age children and adolescents. | 7 months
  Subjects will be given a pre-intervention questionnaire to assess their basic knowledge about influenza infection. Subjects then will play a videogame, designed to be an entertainment-educational hybrid product on influenza infection and influenza vaccination subject. After the intervention, subjects will fill out a post-intervention questionnaire that will assess their knowledge about influenza infection and vaccination.

SECONDARY OUTCOMES:
Increase influenza vaccination in school-age children and adolescents using an entertainment-educational videogame product. | 7 months
  We will assess how many subjects chose to receive the influenza vaccination after playing the educational interactive videogame.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Krilov, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States